CLINICAL TRIAL: NCT03374111
Title: A Multi-center Randomized, Double-blind, Placebo-controlled Study of Colla Corii Asini for the Treatment of Anemia in Pregnant Women With Thalassemia(Presenting the Syndrome of Blood Deficiency)
Brief Title: Colla Corii Asini Treating Anemia in Pregnant Women With Thalassemia(Presenting the Syndrome of Blood Deficiency)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanfang Li, Director, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TH-2
Record Dates: First submitted 2017-12-04; First posted 2017-12-15 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Thalassemia
Keywords: Thalassemia;; the Syndrome of Blood Deficiency; Anemia; Colla Corii Asini
MeSH Terms: conditions — Thalassemia; Anemia | interventions — colla corii asini

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 15g of Colla corii asini granule( produced by Dong-E E-Jiao Co., Ltd) ， taken once daily for 8 weeks
  Interventions: Drug: Colla corii asini
- Control group (Placebo Comparator): a Simulate Agent of Colla corii asini granule， similar in size, shape，color and taste to Colla corii asini granule, taken once daily for 8 weeks
  Interventions: Drug: a Simulate Agent of Colla corii asini granule

INTERVENTIONS:
Drug: Colla corii asini — 15 g Colla corii asini granule daily for 8 weeks
  Other Names: donkey-hide gelatin
  Arms: Experimental group
Drug: a Simulate Agent of Colla corii asini granule — 15 g a Simulate Agent of Colla corii asini granule daily for 8 weeks
  Other Names: Placebo of Colla corii asini granule
  Arms: Control group

SUMMARY:
480 pregnant patients diagnosed of silent or standard α-thalassemia, HbH disease, minor or intermediate β-thalassemia with mild anemia will be randomly assigned to treatment group and control group. Patients in the treatment group will be given 15 g of Colla corii asini powder form daily for 8 weeks and followed up to 42 days postpartum while the control group will be observed and followed up in the same period treated with placebo. Levels of hemoglobin(Hb), reticulocyte (RET), immaturity reticulocyte (IRF), indirect bilirubin(IBIL), total bilirubin(TBIL), lactic dehydrogenase(LDH) will be measured on three visits(baseline, week 4 and week 8). The curative effect of TCM Syndrome( week 8) and undesirable pregnancy outcomes(42 days after giving birth) will be observed.

DETAILED DESCRIPTION:
Thalassemia is a type of hemolytic anemia disease caused by genetic defect of synthesis in one or more globin chains. Among all the single genetic disorders thalassemia has the highest incidence rate in the world and causes heavy burdens on public health system. In China, the southern provinces suffer from high incidence of thalassemia, which is particularly common in the population of Guangdong, Guangxi and Yunnan provinces. Epidemiological studies showed that in Guangdong alone about 17.83 % of the 14,332 pregnant women across 21 regions examined were diagnosed as carriers of thalassemia .

Recent studies showed that compared with healthy controls, women with thalassemia are associated with a wide range of abnormality and adverse pregnancy outcomes including cardiovascular disease, thrombotic disease, spontaneous miscarriage, premature delivery, oligohydramnios, fetal growth restriction and low birth weight. Currently there is no consensus on treating anemia in pregnant thalassemia patients. Due to the absence of an safe and effective therapeutic measures， many thalassemia patients are prone to develop low level of Hb, which can severely impact the fetal growth and maternal health.

In traditional Chinese medicine (TCM), Colla corii asini (CCA, E'jiao) is a gelatin-like traditional Chinese medicine refined from donkey hide and has been widely used in clinical antanemic therapy for more than 2000 years. In the last decade, many studies had addressed the effect of CCA on the anemia using modern pharmacological approaches. The results indicated that CCA contains collagen protein,glycogen and a variety of trace elements, a variety of amino acids, etc. the main components of CCA can promote hematopoiesis by a number of mechanisms which eventually increase the peripheral erythrocyte counts and Hb concentration. Therefore, the investigators proposed that the hematopoietic effects of CCA might also contribute to the treatment of thalassemia with insuffcient or abnormal Hb concentration.

The study aims to evaluate the efficacy and safety of Colla corii asini (CCA ) in improve anemia during pregnancy among silent or standard α-thalassemia, HbH disease, minor or intermediate β-thalassemia. Four hundred and eighty pregnant patients who meet inclusion criteria will be randomly assigned to either the treatment group or control group. Patients in the treatment group will be given 15 g of CCA daily for 8 weeks and followed up to 42 days postpartum, while the control group were observed and followed up in the same period treated with placebo. Levels of hemoglobin (Hb),reticulocyte (RET), immaturity reticulocyte (IRF), indirect bilirubin (IBIL), total bilirubin (TBIL), lactic dehydrogenase (LDH) will be measured on three visits (baseline, week 4 and week 8). The curative effect of TCM Syndrome( week 8) and undesirable pregnancy outcomes(42 days after giving birth) will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed as thalassemia carriers by genetic test with clinical presentation of silent or standard α-thalassemia, HbH disease, minor or intermediate β-thalassemia;
* Patients with mild anemia (70 g/L≤ Hb<100 g/L) prior to study enrollment;
* Singleton pregnancy ;
* Gestational age between 24-32 weeks;
* Patients having not received blood transfusion in the last 12 weeks;
* Written informed consent of the patient.

Exclusion Criteria:

* Known history of allergy or reaction to any component of the investigational product;
* Allergic to two or more drugs;
* Patients with severe thalassemia;
* Anaemia not caused by thalassemia (e.g., iron deficiency, aplastic, megaloblastic or haemolytic anaemia) or bone marrow diseases, leukemia.
* Twin or multiple pregnancies;
* Placental Abnormality (e.g., placenta previa, multilobate placenta, placenta succenturiate, placenta cirumvallate) or polyhydramnios, oligohydramnios, fetal growth restriction, fetal anomaly;
* Patients having received hemopoieticfactors or treated by hematopoietic stem cell transplantation in the last 2 months;
* Hypersplenism or hypertensive disorder in pregnancy;
* Patients with any of the following abnormalities: immunodeficiency, primary diseases involving cardiovascular system, liver, kidney, gastrointestinal tract, endocrine system and hematological system;
* 1.5 times or more higher plasma creatinine level than high limit of normal state;
* 1.5 times or more higher AST or ALT than high limit of normal state;
* Patients with mental illness;
* Patients who suffer from drug or alcohol abuse;
* Patients who addicted to smoking and drinking;
* Participation in any clinical investigational drug study within the previous 3 months;
* Patients who are regarded as ineligible for this study by investigator.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin(Hb) | baseline, week 4 and week 8
  the change of hemoglobin(g/L)

SECONDARY OUTCOMES:
reticulocyte (RET) | baseline, week 4 and week 8
  the change of reticulocyte (RET)count（×10^9/L）
immature reticulocyte fraction（IRF） | baseline, week 4 and week 8
  the change of immature reticulocyte fraction(%)
adverse event | tracked for 42 days after giving birth
  undesirable pregnancy outcomes
indirect bilirubin(IBIL) | baseline, week 4 and week 8
  the change of indirect bilirubin(IBIL)(μmol/L)
total bilirubin(TBIL) | baseline, week 4 and week 8
  the change of total bilirubin(TBIL) (μmol/L)
lactic dehydrogenase(LDH) | baseline, week 4 and week 8
  the change of lactic dehydrogenase(LDH)(U/L)
anaemia cure rates | week 8
  anaemia cure rates(%):The concentration of hemoglobin was higher than baseline > 5g/L;The improvement rate = improved cases/the total number of cases * 100%
The curative effect of TCM Syndrome | week 8
  the change of the TCM syndrome scores of two groups before and after treatment（%）

CONTACTS AND LOCATIONS:
Overall Officials: Yanfang Li, PhD, Principal Investigator — the first affiliated hospital of Guangzhou University of Chinese Medicine ， Guangzhou
Locations (12):
- China (12):
  - The third people's Hospital of Dongguan, Dongguan, Guangdong
  - Intranet of Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - the first affiliated hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Department of Gynaecology and Obstetrics,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Dongguan Guangji Hospital, Guangzhou, Guangdong
  - Shenzhen maternity and child health care hospital, Shenzhen, Guangdong
  - Liuzhou Municipal Matemal and Child Health Hospital, Liuchow, Guangxi
  - The Guangxi Zhuang Autonomous Region National Hospital, Nanning, Guangxi
  - Ruikang Hospital of Guangxi University of Traditional Chinese Medicine, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting in May 2020 when the study have been completed and publication of a clinical trial report.
Access Criteria: the information collected about the study will be used to support other research in the future, and may be shared anonymously with other researchers,data will be freely available to anyone upon request.

REFERENCES:
- [Background] Li Y, He H, Yang L, Li X, Li D, Luo S. Therapeutic effect of Colla corii asini on improving anemia and hemoglobin compositions in pregnant women with thalassemia. Int J Hematol. 2016 Nov;104(5):559-565. doi: 10.1007/s12185-016-2069-0. Epub 2016 Jul 25. PMID 27456464
- [Background] Cheng YL, Zhang XH, Sun YW, Wang WJ, Fang SP, Wu ZK. Clinical Effect and Mechanism of Yisui Shengxue Granules in Thalassemia Patients with Mild, Moderate, or Severe Anemia. Evid Based Complement Alternat Med. 2016;2016:1713897. doi: 10.1155/2016/1713897. Epub 2016 Feb 2. PMID 26949404